CLINICAL TRIAL: NCT01906931
Title: Effective Delivery of Ambulatory Oxygen in Interstitial Lung Disease - a Crossover Trial.
Brief Title: Ambulatory Oxygen for ILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anne Holland (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor-Investigator, Anne Holland, Clinical Chair, Physiotherapy, The Alfred
Organization: The Alfred (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 187_13
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial lung disease; Oxygen therapy; Walk
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Portable Oxygen Concentrator first (Experimental)
  Interventions: Device: Portable oxygen concentrator; Device: Portable oxygen cylinder
- Portable oxygen cylinder first (Active Comparator)
  Interventions: Device: Portable oxygen concentrator; Device: Portable oxygen cylinder

INTERVENTIONS:
Device: Portable oxygen concentrator — Respironics EverGo portable oxygen concentrator on setting 6
  Other Names: Respironics EverGo portable oxygen concentrator
Device: Portable oxygen cylinder — Portable oxygen cylinder at flow rate 5 Litres/min

SUMMARY:
People with interstitial lung disease (ILD) are frequently prescribed ambulatory oxygen, to increase oxygen levels in the blood during daily activities. The best way of delivering this type of oxygen has not been established. The aim of this study is to compare two devices for delivering oxygen in people with interstitial lung disease - the traditional method using portable cylinders and a newer method using a portable concentrator. The investigators hypothesise that oxygen levels during exercise will be significantly higher when using a portable cylinder, but this difference will be small.

DETAILED DESCRIPTION:
Exercise-induced hypoxaemia (EIA) is very common in individuals with ILD, due to progressive lung fibrosis which results in impaired gas exchange. It is common for people with EIA to be prescribed ambulatory oxygen, in order to normalize oxyhaemoglobin saturation, improve oxygen delivery to the tissues and relieve breathlessness during daily activities.

Ambulatory oxygen is traditionally delivered via a refillable portable oxygen cylinder containing compressed gaseous oxygen. More recently, portable oxygen concentrators (POCs) have emerged as a solution to the problem of finite cylinder life and to improve portability. Because a concentrator is constantly extracting oxygen from air, oxygen supply can continue as long as the battery is charged. This is typically around eight hours, but POCs can be recharged from an AC or DC power source. Portable oxygen concentrators usually weigh around 3.5kg, which is significantly lighter than oxygen cylinders, and are much easier to maneuver. However, there are some theoretical disadvantages to POCs. Like all concentrators, they do not deliver 100% oxygen. Concentrations typically range from 85-95%, depending on the flow rate. Differences in pulse timing and peak pulse flow between POCs may affect the fraction of inspired oxygen (FiO2) that is delivered. However, the clinical implications of these differences have not been documented.

The aim of this study is to compare the effects of ambulatory oxygen delivered during exercise using the EverGo POC to ambulatory oxygen delivered with a standard portable cylinder in individuals with ILD. We hypothesise that oxyhaemoglobin saturation during exercise will be significantly higher when using a portable cylinder, but this difference will not be clinically important.

ELIGIBILITY:
Inclusion Criteria:

* a confident diagnosis of ILD made according to established criteria and
* desaturate to less than 90% during a 6-minute walk test

Exclusion Criteria:

* primary diagnosis of a respiratory condition other than ILD (eg COPD)
* currently using continuous oxygen therapy
* oxyhaemoglobin saturation (SpO2) is less than 90% on room air
* unable to perform a 6-minute walk test or comorbidities that limit walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Nadir SpO2 | During 6-min walk test with each oxygen delivery device
  Lowest SpO2 recorded during the 6-min walk test on each device

SECONDARY OUTCOMES:
6-min walk distance | End 6-min walk test with each oxygen delivery device
  The distance walked in 6 minutes with each oxygen delivery device will be compared
Borg dyspnoea score | End 6-min walk test with each oxygen delivery device
  Borg dyspnoea score at the end of the 6-min walk test will be compared between devices
Borg fatigue score | End 6-min walk test with each oxygen delivery device
  Borg fatigue score at the end of the 6-min walk test will be compared between devices
Partial pressure of oxygen in arterial blood (PaO2) at rest | Prior to 6-min walk test with each oxygen delivery device
  PaO2 at rest breathing oxygen from each of the two devices will be compared
Proportion of participants who desaturate to less than 80% | During 6-min walk test on each oxygen delivery device
  Proportion of participants who desaturate to less than 80% with each oxygen delivery device will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia